CLINICAL TRIAL: NCT06534944
Title: The Effect of Nicotinamide Adenine Dinucleotide (NAD) Supplementation on Systemic Vascular Health in Peripheral Artery Disease
Brief Title: NAD Supplementation and Vascular Health in PAD
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15457
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Endothelial function; Cognition
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Pilot open-label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NR supplementation (Experimental): 1g daily NR
  Interventions: Drug: Nicotinamide riboside

INTERVENTIONS:
Drug: Nicotinamide riboside — NR 1g daily for 4 weeks
  Other Names: NR

SUMMARY:
This pilot open-label clinical trial was designed to investigate whether 4-week supplementation with 1g daily NR impacts endothelial function in peripheral circulation, cerebrovascular hemodynamics, cognitive function in older adults with peripheral artery disease.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a prevalent age-related vascular pathology and the third leading cause of cardiovascular morbidity and mortality among older adults. Accumulating evidence indicates that PAD is associated with generalized endothelial dysfunction that expands from the periphery to central circulation and from macro- to microcirculation. One of the mechanisms that contributes to vascular dysfunction in aging and age-related diseases is the decline in the Nicotinamide Adenine Dinucleotide (NAD) levels. Importantly, recent reports indicate that age-associated decreases in NAD are exacerbated in age-related diseases, including in patients with PAD. Clinical data demonstrate that NAD levels can be increased via per os supplementation with the NAD precursor nicotinamide riboside (NR). Although few ongoing studies provide initial evidence that NAD supplementation with NR may benefit vascular health in older adults, including potential improvements in blood pressure and aortic stiffness, the effects of NR supplementation on vascular health in PAD is understudied. This pilot open-label clinical trial was designed to investigate whether 4-week supplementation with 1g daily NR impacts endothelial function in peripheral circulation, cerebrovascular hemodynamics, cognitive function in older adults with peripheral artery disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PAD
* intermittent claudication
* limited walking capacity

Exclusion Criteria:

* macologically uncontrolled type 2 diabetes, hypercholesterolemia, hypertension
* major depressive disorder
* current or prior cerebrovascular complications (including large vessel ischemic stroke with chronic functional impairment)
* neurodegenerative diseases

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in neurovascular coupling using functional near infrared spectroscopy (fNIRS) | 4 weeks
  Functional near infrared spectroscopy (fNIRS) will be performed during the cognitive n-back task. fNIRS approach generates data that represent a relative change in oxygenated and deoxygenated hemoglobin measured over the cortical brain tissues. Neurovascular coupling will be evaluated as a change in oxy- and deoxy-hemoglobin between before and after treatment. Units of measure - beta. Reported as a change from baseline, before and after treatment.
Change in macrovascular endothelial function | 4 weeks
  Changes in macrovascular endothelial function will be assessed using sonography during flow mediated dilation approach. The change in brachial artery diameter (mm) is calculated and reported as a %change from baseline, between before and after treatment.
Change in Attention | 4 weeks
  The allocation of one's limited capacities to deal with an abundance of environmental stimulation will be measured in a combined "Flanker Inhibitory Control and Attention Test".Units of measure - score (from 0 to 10, bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Episodic Memory | 4 weeks
  Cognitive processes involved in the acquisition, storage and retrieval of new information, will be measured using the "Picture Sequence Memory Test". Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Working Memory | 4 weeks
  The ability to store information until the amount of information to be stored exceeds one's capacity to hold that information will be measured using the "List Sorting Working Memory Test". Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Language | 4 weeks
  Picture Vocabulary Test measures receptive vocabulary administered in a computer-adaptive test (CAT) format. Respondents select the picture that most closely matches the meaning of the word, before and after treatment. Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Executive Function | 4 weeks
  The capacity to plan, organize and monitor the executive of behaviors that are strategically directed in a goal-oriented manner will be measured using the "Dimensional Change Card Sort Test". Units of measure - score (from 0 to 10, bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Processing Speed | 4 weeks
  Pattern Comparison Processing Speed Test assesses the amount of information that can be processed within a certain unit of time. Items are simple so as to purely measure processing speed. Units of measure - score (from 0 to 130, bigger number is better). Reported as a %change from baseline, before and after treatment.
Blood collection | 4 weeks
  Blood samples will be used in in vitro assays to measure the effect of treatment on endothelial function.
Change in microvascular endothelial function | 4 weeks
  Changes in microvascular endothelial function will be assessed using laser speckle contrast imaging (LSCI) in the hand using the flow mediated dilation approach. The change in skin perfusion is calculated and reported as a %change from baseline, between before and after treatment. Units of measure - perfusion index (arbitrary units). Reported as a baseline and maximal perfusion, arbitrary units

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified data, including participants age, sex, diagnosis, as well as experimental evaluation data will be shared with researchers via publication in the scientific journals and/or biomedical online repositories
Supporting Information: Study Protocol, SAP